CLINICAL TRIAL: NCT04289337
Title: Double-blind Clinical Trials of Probiotic Products in Oral Health.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glac Biotech Co., Ltd (Industry)
Responsible Party: Principal Investigator, Hsieh-Hsun Ho, R.D. Manager Doctor, Glac Biotech Co., Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CS19052
Record Dates: First submitted 2020-02-24; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Probiotics; Oral Health; Probiotic Metabolites

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Combined probiotics (1) (Experimental): Combined Lactobacillus salivarius subsp. salicinius AP-32, Bifidobacterium animalis subsp. lactis CP-9 and Lactobacillus paracasei ET-66.
  Interventions: Dietary Supplement: Combined probiotics (1)
- Combined probiotics (2) (Experimental): Combined Lactobacillus salivarius subsp. salicinius AP-32, Lactobacillus plantarum LPL28 and Lactobacillus paracasei ET-66.
  Interventions: Dietary Supplement: Combined probiotics (2)
- Combined heat-killed probiotics (1) (Experimental): Combined heat-killed Lactobacillus salivarius subsp. salicinius AP-32, Bifidobacterium animalis subsp. lactis CP-9 and Lactobacillus paracasei ET-66.
  Interventions: Dietary Supplement: Combined heat-killed probiotics (1)
- Combined heat-killed probiotics (2) (Experimental): Combined heat-killed Lactobacillus salivarius subsp. salicinius AP-32 and Lactobacillus paracasei ET-66.
  Interventions: Dietary Supplement: Combined heat-killed probiotics (2)
- Probiotic metabolites (Experimental): Combined Lactobacillus salivarius subsp. salicinius AP-32, Lactobacillus plantarum LPL28 and Lactobacillus paracasei ET-66 metabolites.
  Interventions: Dietary Supplement: Probiotic metabolites
- Placebo (Placebo Comparator): Does not contain probiotics, heat-killed probiotics and related metabolites.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Combined probiotics (1) — Subjects used one oral combined probiotics (1) tablet each morning, noon, and evening for 4 weeks.
  Arms: Combined probiotics (1)
Dietary Supplement: Combined probiotics (2) — Subjects used one oral combined probiotics (2) tablet each morning, noon, and evening for 4 weeks.
  Arms: Combined probiotics (2)
Dietary Supplement: Combined heat-killed probiotics (1) — Subjects used one oral combined heat-killed probiotics (1) tablet each morning, noon, and evening for 4 weeks.
  Arms: Combined heat-killed probiotics (1)
Dietary Supplement: Combined heat-killed probiotics (2) — Subjects used one oral combined heat-killed probiotics (2) tablet each morning, noon, and evening for 4 weeks.
  Arms: Combined heat-killed probiotics (2)
Dietary Supplement: Probiotic metabolites — Subjects used one oral probiotic metabolites tablet each morning, noon, and evening for 4 weeks.
  Arms: Probiotic metabolites
Dietary Supplement: Placebo — Subjects used one oral placebo tablet each morning, noon, and evening for 4 weeks.
  Arms: Placebo

SUMMARY:
In order to evaluate the effects of supplementary probiotics and their metabolites on oral environment and oral microbiota, Taiwan FDA No. 88037803 will be used to evaluate the effects of oral probiotic candidate strains from previous research results and develop oral probiotic products.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 20 to 40 years old.
* More than 10^5 Streptococcus mutans (CFU/mL) of saliva.

Exclusion Criteria:

* Smoking.
* Subject has major illness.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
The change from baseline colony-forming unit (CFU) of Streptococcus mutans at 4 weeks. | 4 weeks.
  The plaque on the inside and outside of teeth was collected by cotton swab and putting in the microbial culture broth before and after taking the oral tablets. The microbial culture broth will be diluted and smeared on the mitis salivarius-bacitracin agar (MSBA) plate for counting the CFU of Streptococcus mutans.
The change from baseline concentration of saliva immunoglobulin A (IgA) at 4 weeks. | 4 weeks.
  The saliva was collected by the centrifuge tube before and after taking the oral tablets. IgA will be detected by enzyme-linked immunosorbent assay (ELISA).
The change from baseline microbiota at 4 weeks. | 4 weeks.
  The saliva was collected by the next-generation sequencing (NGS) saliva collection tube before and after taking the oral tablets. The changes in microbial flora will be detected by NGS.

SECONDARY OUTCOMES:
The change from baseline CFU of total oral microbiota at 4 weeks. | 4 weeks.
  The plaque on the inside and outside of teeth was collected by cotton swab and putting in the microbial culture broth before and after taking the oral tablets. The microbial culture broth will be diluted and smeared on the plate count agar (PCA) plate for counting the CFU of total oral microbiota.
The change from baseline CFU of probiotics at 4 weeks. | 4 weeks.
  The plaque on the inside and outside of teeth was collected by cotton swab and putting in the microbial culture broth before and after taking the oral tablets. The microbial culture broth will be diluted and smeared on the De Man, Rogosa and Sharpe agar (MRSA) plate for counting the CFU of probiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Hsieh-Hsun Ho, Ph.D., Principal Investigator — Glac Biotech Co., Ltd
Locations (1):
- Glac Biotech Co., Ltd, Tainan, Taiwan